CLINICAL TRIAL: NCT01651091
Title: Effects of Meditation Awareness Training on Psychosocial Functioning in Prison Participants: A Randomized Controlled Trial
Brief Title: Effects of Meditation Awareness Training on Psychosocial Functioning in Prison Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham Trent University (Other)
Collaborators: Awake to Wisdom Foundation (Unknown); Serco Group Plc (Unknown)
Responsible Party: Principal Investigator, Edo Shonin, Research Psychologist, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MAT-30072012-T
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Psychosocial Functioning
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation Awareness Training (Experimental)
  Interventions: Other: Meditation Awareness Training
- Treatment as Usual (Active Comparator)
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Meditation Awareness Training — Psychotherapy Intervention
  Arms: Meditation Awareness Training
Other: Treatment as usual
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to investigate the effects of an eight-week long group-based secular intervention known as Meditation Awareness Training (MAT) on psychosocial functioning in prison participants.

DETAILED DESCRIPTION:
In Western practitioner settings, Buddhist principles are increasingly being used in the treatment of a wide range of mental health issues. However, there is a dearth of high quality research examining the effects of Buddhist-derived interventions (BDIs) on mental health in forensic settings. The purpose of this study is to assess the salutary effects and acceptability of a secularised group-based eight-week BDI known as Meditation Awareness Training (MAT) against relevant predictors of adaptive psychosocial functioning and mental health in violent offenders. A randomized controlled trial (RCT) design will be employed structured with reference to CONSORT (Consolidated Standards of Reporting Trials) 2010 guidelines. English speaking adult males (aged 18-65 years) serving indeterminate prison sentences for offences of instrumental violence at a category B prison will be invited to receive MAT on a voluntary basis. Computer-generated numbers will be used to randomly allocate prison participants (n=102 - based on statistical power calculations) to either an intervention or 'treatment as usual' (TAU) control condition. Measures will be taken pre- and post-intervention and at three-month follow-up to assess maintenance effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult male (aged 18 to 65)
* English speaking
* Intact cognition(mini-mental status exam ≥23)
* Incarceration for an act of instrumental violence
* Evidence of self-harming and/or suicidal ideations and/or substance-use during the 12 months prior to the study.

Exclusion Criteria:

* current participation in a program of structured psychotherapy or counselling
* any prior formal meditation training
* psychopharmacology commenced or dosage changed one-month prior to intervention (stable medication permitted)

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Risk of Reoffending

SECONDARY OUTCOMES:
Anger levels
Self-esteem
Substance-use locus of control
Self-harming
Affective mood states

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, United Kingdom